CLINICAL TRIAL: NCT02361554
Title: Deep Brain Stimulation in Treatment Resistant Schizophrenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00042065; 1U01MH130625-01A1 (NIH)
Record Dates: First submitted 2015-02-06; First posted 2015-02-11 (Estimated); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Treatment-resistant Schizophrenia
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Deep Brain Stimulation Implant (Experimental): Unblinded treatment arm, deep brain stimulation of the substantia nigra pars reticulata for treatment resistant schizophrenia.
  Interventions: Device: Medtronic Percept with SensSight Deep Brain Stimulation System

INTERVENTIONS:
Device: Medtronic Percept with SensSight Deep Brain Stimulation System — Placement of Deep brain stimulation System for treatment of chronic auditory hallucinations in treatment-resistant schizophrenia

SUMMARY:
The purpose of this pilot study is to investigate the use of deep brain stimulation (DBS) of the substantia nigra pars reticulata (SNr) in subjects with treatment-resistant schizophrenia. There is a subset of patients with schizophrenia who continue to have persistent psychotic symptoms (auditory hallucinations and delusions) despite multiple adequate medication trials with antipsychotic medications including clozapine. There are currently no available treatments for such patients who generally have poor function and are chronically disabled, unable to work, live independently or have meaningful social relationships. Neuroimaging studies in patients with schizophrenia have revealed information about pathological neural circuits that could be suitable targets using deep brain stimulation. Although not yet tested in patients with schizophrenia, DBS is in early phase clinical trials in other psychiatric disorders.

This pilot study will investigate the use of DBS in treatment-resistant schizophrenia subjects who have exhausted all other therapeutic alternatives but continue to have persistent disabling psychotic symptoms. Of note, DBS is not FDA approved for use in patients with schizophrenia. The method will be similar to that used in subthalamic nucleus stimulation in patients with Parkinson's Disease. However, the electrode will be advanced slightly inferior into the SNr, a major outflow nucleus of the basal ganglia, with the intention of causing local inhibition of SNr outflow resulting in disinhibition of the mediodorsal nucleus (MDN) of the thalamus. Hypofunction of the MDN has been implicated in the pathophysiology of schizophrenia in post-mortem as well as multiple structural and functional imaging studies. Evidence suggests that dysfunction of the MD is implicated in both positive and cognitive symptoms (such as working memory impairment) in schizophrenia. Frequent monitoring and clinical assessment with psychiatric scales will be used to monitor treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Males and females who are at least 22 years of age.
* Subject has a diagnosis of schizophrenia or schizoaffective disorder as determined by a review of medical records, discussion with referring psychiatrist as well as the Structured Clinical Interview for DSM-V (SCID-V).
* Subject determined to be treatment-resistant for at least one year prior to the Screening Visit as demonstrated by clinical evidence (determined by review of medical records and discussion with referring psychiatrist) of persistent auditory hallucinations and/or delusions that have not responded to treatment with three adequate regimens of antipsychotic medication including one failed trial of clozapine as defined as follows:

  1. Adequate trials of two different antipsychotic drugs (not including clozapine) belonging to different classes of at least 12 weeks equivalent to at least 500 mg/day of chlorpromazine within the previous 5 years.
  2. A trial of clozapine of at least12 weeks at a dose of at least 400 mg (or a clozapine level of at least 350 ng/mL). Subjects who were unable to tolerate clozapine at this dose or for this duration because of intolerable side effects are also eligible.
* Subject has at least a score of 6 (severe) on 2 of the 4 BPRS positive symptoms (conceptual disorganization, grandiosity, hallucinatory behavior and unusual thought content) at all three Baseline Visits prior to undergoing surgery. One of the 2 must be hallucinatory behavior.
* Subject must be ambulatory.
* Females who are postmenopausal, physically incapable of childbearing, or practicing an acceptable method of birth control. Acceptable methods of birth control include surgical sterilization, hormonal contraceptives, or double-barrier methods (condom or diaphragm with a spermicidal agent or intrauterine device [IUD]). If practicing an acceptable method of birth control, a negative urine pregnancy test result has been obtained at baseline Visits 1 and 3.
* Subject is determined by independent psychiatrist with expertise in capacity assessments to have decision-making capacity to provide informed consent.
* Subject is able to read English, understand and cooperate with study procedures, and has signed a written informed consent form prior to any study procedures.

Exclusion Criteria:

* Subject has a positive urine drug screen at any of the three Baseline Visits.
* Subject had major surgery within three months prior to Baseline Visit 1 or has other surgery planned during the proposed study period.
* Subject is determined by medical consultant to have medical contraindications to undergoing surgery.
* Subject is pregnant or breast-feeding.
* Subject has a history of alcohol or drug abuse within the past 6 months and dependence within the past year.
* Subject has a medical illness/condition, co-morbid psychiatric illness, and/or abnormal diagnostic finding that would interfere with the completion of the study, confound the results of the study, or pose risk to the patient.
* Subject has participated in another investigational drug trial or therapeutic trial within 30 days of Baseline Visit 1.
* Subject has a diagnosis of mental retardation.
* Subject has a neurological condition, or a history of traumatic brain injury associated with loss of consciousness of > 1 hour and/or intracranial/epidural/subdural bleeding.
* Subject has defibrillator or pacemaker or other implants that will interfere with MRI and functioning of the device.
* Unstable psycho-social condition including housing and poor support.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Brief Psychiatric Rating Scale | 1 year after neurostimulator implantation
  We will assess deep brain stimulation effects on the positive and psychosis features of schizophrenia.
Change from baseline in the Scales for the Assessment of Negative Symptoms (SANS) | 1 year after neurostimulator implantation
  We will assess deep brain stimulation effects on negative symptoms aspects of schizophrenia.
Incidence of adverse device effects (ADEs). | 1 year after neurostimulator implantation
  We will assess the incidence of adverse device effects as defined by the Code of Federal Regulations (21 CFR 812.3)

SECONDARY OUTCOMES:
Change from baseline in the Young Mania scale (YMS) | 1 year after neurostimulator implantation
  We will assess deep brain stimulation effects on mania as assessed by the YMS.
Change from baseline in the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) cognitive test battery. | 1 year after neurostimulator implantation
  We will assess deep brain stimulation effects on cognition as assessed by the MATRICS cognitive test battery.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Cascella, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States